CLINICAL TRIAL: NCT03391895
Title: The Effect of the Inspiratory Muscle Training on Respiratory Muscle Strength, Respiratory Function and Functional Capacity in Adolescents With Idiopathic Scoliosis
Brief Title: The Effect of the Inspiratory Muscle Training on Respiratory Parameters and Functional Capacity in Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Gözde Başbuğ, Lecturer, PT, MSc, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BVUgbasbug01
Record Dates: First submitted 2017-12-29; First posted 2018-01-05 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent Idiopathic Scoliosis; Scoliosis; Inspiratory Muscle Training; Exercise Training; Respiratory Exercise Training; Pulmonary Function Test; 6-Minute Walk test; Respiratory Muscle Strength
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients in this group will receive a home based exercise program. Home based exercise program includes deep diaphragmatic breathing exercises, resistive local expansion exercise on the collapsed areas in scoliosis concave sides, dynamic lumber stabilization, strengthening of inter scapular muscles, posture and stretching exercises once a day for 8 weeks. One of the exercise sessions was supervised by physiotherapist each week.
  Interventions: Other: Home based exercise program
- Training Group (Experimental): In addition to home based exercise program, patients in this group will also receive inspiratory muscle training for 15 minutes, twice a day, 7 days a week for 8 weeks. One exercise session will be supervised in our clinic per week, other sessions will be performed at home.
  Interventions: Other: Home based exercise program; Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Home based exercise program — Program will include deep diaphragmatic breathing exercises, local expansion exercise on the collapsed areas in scoliosis concave sides with elastic exercise bands, dynamic lumber stabilization exercises for core stabilisation, strengthening of interscapular muscles with elastic bands and stretching exercises for lumbar extensor, hip flexor and hamstring muscles. Exercises will be applied 2 sets of 10 repetitions and once a day.
Other: Inspiratory Muscle Training — Threshold IMT device will be used for the training. Training intensity will set at 30% of the maximum inspiratory pressure after assessment of respiratory muscle strength for each patient every week.
  Arms: Training Group

SUMMARY:
Scoliosis is the abnormality of the spine with direct effects on the shape and mechanics of the thoracic cage. Adolescent Idiopathic Scoliosis (AIS) is the most common 3-dimensional deformity of the spine which can potentially affect respiratory function, exercise capacity as well as the performance of inspiratory and expiratory muscles. During growth morphological changes of thoracic cage affects the pulmonary tissues and functions. Respiratory functions shows negative changes due to Cobb angle, curve localization, number of vertebra and onset age in patient with scoliosis.

Exercise approaches include respiratory training program and aim to improve respiratory functions.It is reported that respiratory muscle weakness is a potent contributor to pulmonary impairment in mild, moderate, and severe forms of scoliosis. Studies showed that exercise training and respiratory exercises may improve respiratory function and exercise capacity in patients with AIS. Thus the aim of this study was to investigate the effect of inspiratory muscle training on respiratory muscle strength, respiratory function and functional capacity in adolescents with idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent Idiopathic Scoliosis diagnosis

Exclusion Criteria:

* Documented diagnosis any of cardiopulmonary, neurological, orthopedic or mental disorders which may affect the assessment results.
* Subjects previously involved in exercise training or physiotherapy programs
* Subjects previously undertaken any of spinal surgeries.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline Forced Vital Capacity (FVC) at 8 weeks | Eight weeks
Change from baseline Forced Expiratory Volume in 1 second (FEV1) at 8 weeks | Eight weeks
Change from baseline Peak Expiratory Flow (PEF) at 8 weeks | Eight weeks
Change from baseline Maximum Inspiratory Pressure (MIP) at 8 weeks | Eight weeks
Change from baseline Maximum Expiratory Pressure (MEP) at 8 weeks | Eight weeks
Change from baseline distance covered in six-minute walk test at 8 weeks | Eight weeks

SECONDARY OUTCOMES:
Change from baseline thoracic axial trunk rotation (ATR) | Eight weeks
  Measurements will be applied with Bunnell Scoliometer by a qualified physiotherapist.
Change from baseline thoracic-lumber junction axial trunk rotation (ATR) | Eight weeks
  Measurements will be applied with Bunnell Scoliometer by a qualified physiotherapist.
Change from baseline lumber axial trunk rotation (ATR) | Eight weeks
  Measurements will be applied with Bunnell Scoliometer by a qualified physiotherapist.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided